CLINICAL TRIAL: NCT05822934
Title: Carboplatin-gemcitabine Versus Cisplatin-gemcitabine as Neoadjuvant Chemotherapy for Treatment of Muscle Invasive Urinary Bladder Cancer: a Prospective Randomized Trial
Brief Title: Carboplatin-gemcitabine Versus Cisplatin- Gemcitabine as Neoadjuvant Chemotherapy for Treatment of Muscle Invasive Urinary Bladder Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Mahmoud Moustafa Abdelakher, Doctor principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Urinary bladder cancer
Record Dates: First submitted 2023-01-24; First posted 2023-04-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Urinary Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carboplatin-gemcitabine (Experimental): 3-4 cycles of Carboplatin-Gemcitabine as a neoadjuvant treatment for Urinary bladder cancer Muscle invasive
  Interventions: Drug: Carboplatin-Gemcitabine Cisplatin-Gemcitabine
- cisplatin-gemcitabine (Active Comparator): 3-4 cycles of Cisplatin -Gemcitabine as a neoadjuvant treatment for Urinary bladder cancer Muscle invasive
  Interventions: Drug: Carboplatin-Gemcitabine Cisplatin-Gemcitabine

INTERVENTIONS:
Drug: Carboplatin-Gemcitabine Cisplatin-Gemcitabine — Carboplatin-gemcitabine versus cisplatin-gemcitabine as neoadjuvant chemotherapy for treatment of muscle invasive urinary bladder cancer

SUMMARY:
Patients will be randomized in 1:1 ratio to two treatment groups first group will receive 3-4 cycles of neoadjuvant Carboplatin(AUC4)-Gemcitabine (treatment group) and second group will receive 3-4 cycles of neoadjuvant Cisplatin(75mg/m2 Day1)-Gemcitabine (Control group). Patients will undergo radiological assessment, full laboratory work up, and cystoscopy before undergoing either radical cystectomy or Definitive Radiotherapy concurrent with chemotherapy

DETAILED DESCRIPTION:
Patients will be randomized in 1:1 ratio to two treatment groups first group will receive 3-4 cycles of neoadjuvant Carboplatin(AUC4)-Gemcitabine (treatment group) and second group will receive 3-4 cycles of neoadjuvant Cisplatin(75mg/m2 Day1)-Gemcitabine (Control group). Patients will undergo radiological assessment, full laboratory work up, and cystoscopy before undergoing either radical cystectomy or Definitive Radiotherapy concurrent with chemotherapy. After finishing treatment, all patients should undergo follow up every 3 months for two years then six monthly thereafter .Follow up will include History, physical examination, full laboratory works (CBC, renal function testing and liver function testing). Imaging by CT or MRI abdomen and pelvis for all patients and cystoscopy in bladder preservation protocol

ELIGIBILITY:
Inclusion Criteria:All patients diagnosed with muscle invasive urinary bladder cancer that can receive chemotherapy are included the criteria are

* • Age above 18 years,

  * Pathologically proven urinary bladder cancer,
  * Patients with clinical stages T2-4a N0-3 M0,
  * Patients with good renal and liver functions
  * patients with no distant metastases,
  * no other malignancy (double malignancy).
  * Performance status 0-1 according to ECOG performance status scale.
  * Patients with no contraindications for radiotherapy.

Exclusion Criteria:

* • performance status 2-4 according to ECOG performance status scale.

  * patients refuse to receive chemotherapy,
  * patients not eligible to receive chemotherapy due to liver or renal impairment or thrombocytopenia,
  * patients with M1 disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt